CLINICAL TRIAL: NCT03095118
Title: Single-center Phase 2 Open-label Trial Evaluating Efficacy and Safety of Daratumumab in Treatment of Patients With Proliferative Glomerulonephritis With Monoclonal Immune Deposits and C3 Glomerulopathy Associated With Monoclonal Gammopathy
Brief Title: Daratumumab in Treatment of PGNMID and C3 GN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fernando Fervenza (Other)
Responsible Party: Sponsor-Investigator, Fernando Fervenza, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-004805
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Results first posted 2021-07-16 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Membranoproliferative Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab (Experimental): Subjects will receive daratumumab intravenously at a dose of 16 mg/kg once weekly for 8 weeks followed by once every 2 weeks for 8 additional doses
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Intravenously (IV) at a dose of 16 mg/kg once weekly for 8 weeks, followed by once every 2 weeks for eight additional doses
  Other Names: Darzalex

SUMMARY:
This study is being done to see if daratumumab is safe and effective in the treatment of proliferative glomerulonephritis with monoclonal immune deposits (PGNMID) and C3 glomerulopathy associated with monoclonal gammopathy (C3GN). This is an inflammatory disease in the kidney due to the production of abnormal proteins. There are no known standard effective treatments for patients with PGNMID and C3GN secondary to monoclonal gammopathy. These diseases are caused by abnormal production of proteins (monoclonals) by abnormal clones. Daratumamb has been shown to be effective in treating patients with multiple myeloma a disease which also caused by over production of monoclonal proteins from abnormal clones. Everyone in this study will receive daratumumab.

DETAILED DESCRIPTION:
This study is an open-label phase 2 trial of the safety and efficacy of daratumumab, in the treatment of PGNMID and C3GN associated with monoclonal gammopathy. Subjects will be screened at outpatient Nephrology Clinic visit appointments and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained baseline values will be established and subjects will begin treatment and follow-up for the next 12 months. Daratumumab will be administered once weekly for 8 weeks and then once every 2 weeks for 8 additional doses. Patients will be followed for a total of 12 months (6 months after the last infusion). A final visit for evaluation and collection of lab samples will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Renal biopsy read at Mayo Clinic confirming the diagnosis of PGNMID or C3 GN
* In cases of C3GN serum electrophoresis with immunofixation should confirm presence of monoclonal gammopathy
* Proteinuria ≥ 1000 mg over 24 hours
* eGFR ≥ 20 mL/min/SA
* Subjects able and willing to give informed consent

Exclusion Criteria:

* Pregnancy
* Hepatitis B or C, HIV
* Multiple myeloma
* Anemia with Hgb < 8.5 g/dL
* Thrombocytopenia with platelet count < 100,000
* Leukopenia with WBC < 3.5
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication
* Unable to provide consent
* Patients receiving therapy with oral prednisone or glucocorticoid equivalent in the last 6 weeks
* Patients who had received immunosuppressive therapy including cyclophosphamide, MMF, cyclosporine, tacrolimus or azathioprine in the last 3 months
* Patients who received rituximab previously with CD20 count of zero at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C Fervenza, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Zand L, Rajkumar SV, Leung N, Sethi S, El Ters M, Fervenza FC. Safety and Efficacy of Daratumumab in Patients with Proliferative GN with Monoclonal Immunoglobulin Deposits. J Am Soc Nephrol. 2021 May 3;32(5):1163-1173. doi: 10.1681/ASN.2020101541. Epub 2021 Mar 8. PMID 33685975
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daratumumab
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Diagnosis not associated with monoclonal gammopathy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daratumumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (20.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events
Description: Number of treatment-emergent adverse events as defined as major infection (defined as the development of pneumonia, severe urinary tract infection/pyelonephritis, sepsis, meningitis), grade 3 or 4 anemia, leukopenia, or thrombocytopenia.
Time Frame: 1 year
Measure: Number; unit: Serious Adverse Events
Arm/Group | Daratumumab
Number analyzed (Participants) | 12
Serious Adverse Events | 5

2. Secondary Outcome: Remission Status at 6 Months
Description: The number of subjects to reach either complete remission or partial remission at 6 months after infusion.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
Participants | 8

3. Secondary Outcome: Remission Status at 12 Months
Description: The number of subjects to reach either complete remission or partial remission at 12 months after infusion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
Participants | 9

4. Secondary Outcome: Proteinuria at Baseline
Description: Measured using 24 hour urine collection reported in mg/24h
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: mg/24h
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
mg/24h | 4346 [3245 to 7943]

5. Secondary Outcome: Proteinuria at 6 Months
Description: Measured using 24 hour urine collection reported in mg/24 h
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/24h
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
mg/24h | 702 [435 to 3057]
Statistical Analysis 1: Comparison: Daratumumab; Proteinuria baseline values compared to 6 month follow up values; Test type: Superiority; p = 0.001, t-test, 2 sided

6. Secondary Outcome: Proteinuria at 12 Months
Description: Measured using 24 hour urine collection reported in mg/24h
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: mg/24h
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
mg/24h | 1264 [463 to 3645]
Statistical Analysis 1: Comparison: Daratumumab; Proteinuria baseline values compared to 12 month follow up values; Test type: Superiority; p = 0.004, t-test, 2 sided

7. Secondary Outcome: Serum Creatinine at Baseline
Description: Blood serum collected and reported in mg/dL
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
mg/dL | 1.36 (0.57)

8. Secondary Outcome: Serum Creatinine at 6 Months
Description: Blood serum collected and reported in mg/dL
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
mg/dL | 1.25 (0.44)
Statistical Analysis 1: Comparison: Daratumumab; Serum creatinine baseline values compared to 6 month follow up values; Test type: Superiority; p = 0.15, t-test, 2 sided

9. Secondary Outcome: Serum Creatinine at 12 Months
Description: Blood serum collected and reported in mg/dL
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Daratumumab
Number analyzed (Participants) | 10
mg/dL | 1.25 (0.52)
Statistical Analysis 1: Comparison: Daratumumab; Serum creatinine baseline values comparted to 12 month follow up values; Test type: Superiority; p = 0.16, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 1 year on all participants.
Arm/Group | Daratumumab
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab (N=12)
Eye Chemosis (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Acute Glaucoma (Eye disorders) | 1 (1)
Fever (General disorders) | 1 (1)
C. difficile infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab (N=12)
UTI (Renal and urinary disorders) | 2 (2)
URI (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (16)
Congestion (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Throat Irritation (General disorders) | 6 (11)
Blurred Vision (Eye disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Tingling in feet (General disorders) | 3 (4)
Flushed (General disorders) | 2 (3)
Watery eyes (Eye disorders) | 2 (2)
Itching (General disorders) | 2 (3)
Sneezing (General disorders) | 1 (1)
Chest tightness (General disorders) | 1 (1)
Vagal response (Cardiac disorders) | 1 (1)
Lip tingling (General disorders) | 1 (2)
Skin itchy at IV site (Skin and subcutaneous tissue disorders) | 1 (2)
Hoarse voice (General disorders) | 1 (1)
Sensation of facial swelling (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Nausea (General disorders) | 2 (2)
Insomnia (General disorders) | 1 (2)
Night sweats (General disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Sore throat (General disorders) | 2 (2)
Leg cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Sore scalp (Skin and subcutaneous tissue disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Restless legs (Nervous system disorders) | 1 (1)
Sore in mouth (General disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Foot pain (General disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT03095118/Prot_SAP_000.pdf